CLINICAL TRIAL: NCT06900985
Title: Assessment of a Psychological Treatment for Smoking Cessation Combined With an App According to the Intensity of Therapeutic Contact: Randomized Controlled Trial
Brief Title: Therapeutic Contact Intensity in a Psychological Smoking Cessation Intervention With an App
Acronym: TREATINTSMOKE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Ana López Durán, Phd in Clinical Psychology and Psychobiology/Associated Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID2023-146663OB-I00
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Smoking Behaviors
Keywords: smoking; treatment; cognitive-behavioral; therapeutic-contact intensity; digital intervention; eHealth; randomized controlled trial
MeSH Terms: conditions — Smoking | interventions — Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1. High-intensity therapeutic contact cognitive-behavioral treatment for smoking cessation with App (Active Comparator): It will consist of an App and 8 one-hour sessions applied in group format once a week (8 weeks total duration). The sessions will be conducted by trained clinical psychology/general health psychology professionals and will be carried out using video calls.
  Interventions: Behavioral: 8-sessions CBT + App
- 2. Medium-intensity therapeutic contact CBT for smoking cessation with App (Active Comparator): It will consist of an App and 4 one-hour sessions applied in group format every two-weeks (8 weeks total duration). The sessions will be conducted by trained clinical psychology/general health psychology professionals and will be carried out using video calls.
  Interventions: Behavioral: 4-sessions CBT+App
- 3. App only (no therapeutic-contact group). (Active Comparator): It will consist of the same App than participants assigned to Conditions 1 and 2, but without contact with professionals
  Interventions: Behavioral: Smoking cessation App

INTERVENTIONS:
Behavioral: 8-sessions CBT + App — It will consist of 8 one-hour sessions applied in group format once a week and participants will be followed at 3, 6, and 12 months. The sessions will be conducted by clinical psychology/general health psychology professionals and will be carried out using video calls. The smoking cessation treatment follows a cognitive-behavioral approach with components for anhedonia reduction, increased physical activity and positive social support, being a modified, multidisciplinary, and extended version of the original smoking cessation program (Becoña, 2007; Becoña et al., 2017). The treatment will be complemented with an App with active therapeutic components that participants will use during treatment and the one-year follow-up period.
  Arms: 1. High-intensity therapeutic contact cognitive-behavioral treatment for smoking cessation with App
Behavioral: 4-sessions CBT+App — It will consist of 4 one-hour sessions applied in group format every two-weeks (8 weeks total duration) and participants will be followed at 3, 6, and 12 months. The sessions will be conducted by clinical psychology/general health psychology professionals and will be carried out using video calls. The 4 sessions will have the following content: 1) explanation of treatment rationale and components available in the App; 2) participants' progress monitoring, reinforcement of achieved goals, and analysis of difficulties; 3) cessation planning support; and 4) relapse prevention support. The treatment sessions will be protocolized in a treatment manual. The treatment will be complemented with the same App that the other conditions
  Arms: 2. Medium-intensity therapeutic contact CBT for smoking cessation with App
Behavioral: Smoking cessation App — It will consist in the same App than the other two conditions. No therapeutic contact will be avaliable.
  Arms: 3. App only (no therapeutic-contact group).

SUMMARY:
This randomized controlled trial intends to examine the efficacy of a smoking cessation intervention with an App according to the intensity of therapeutic contact. Participants will be assigned to one of three groups. The first group will receive eight sessions with trained psychologists alongside access to the App. The second group will receive four sessions with trained psychologists plus App access. The control group will only have access to the App. This study seeks to determine the impact of different levels of therapeutic contact on abstinence outcomes.

DETAILED DESCRIPTION:
Smoking remains the leading preventable cause of morbidity and mortality worldwide. It is crucial to implement preventive measures to reduce the likelihood of people starting to smoke but also to make effective smoking cessation treatments available to those who smoke. Psychological interventions have proven to be effective to quit smoking and are considered first-choice interventions, especially for specific populations such as adolescents or pregnant women . The motivation behind this proposal is to improve the effectiveness of smoking cessation treatments based on our clinical and research experience in smoking cessation psychological interventions. Although we have very effective psychological treatments, producing abstinence rates of approximately 70% at the end of the treatment, and 35% at one year of follow-up to continue improving its effectiveness and reduce relapse rates is warranted. Furthermore, technological advances can help increase accessibility to available treatments and motivation to participate in smoking cessation interventions.

The main objective of this proposal is to assess the efficacy of a cognitive-behavioral treatment for smoking cessation with new components (anhedonia and mood management, physical activity, and positive social support) according to the intensity of the therapeutic contact, through a randomized controlled trial. The treatment will be conducted through video call format to make it more accessible. The study will compare three groups that will receive treatments of varying intensity of therapeutic contact: 1) 8 intervention sessions + App (Experimental Group 1, EG1), 2) 4 intervention sessions + App (Experimental Group 2, G2), and 3) no therapeutic contact, App only (control group/CG). Our initial hypothesis is that the higher intensity intervention (EG1) will be more effective than EG2 and CG groups in abstinence outcomes at the end of the intervention and in reducing relapse rates for one year follow-up. The EG2 will be more effective than the CG in abstinence outcomes at the end of the intervention and in reducing relapse rates during one-year follow-up.

Digital treatment delivery formats will be used to increase treatment accessibility: 1) treatment sessions will be conducted through video calls which will remove geographical and time-related barriers. This format will be particularly useful for smokers experiencing barriers to access to treatment due to work/family schedules; 2) a smoking cessation App will be used to improve adherence and access to treatment components anytime, anywhere. Moreover, integrating technology into the treatment can facilitate participants intersessions tasks and support the work of professionals. Our previous experience with an App as a complement to the smoking cessation intervention showed excellent abstinence outcomes.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or over
* wishing to participate in the treatment
* providing written informed consent
* smoking at least 5 cigarettes per day
* completion of all pre-treatment assessment questionnaires
* having a valid email address
* having an Android or iOS smartphone and being willing to use it throughout the treatment

Exclusion Criteria:

* a diagnosis of severe mental disorder (bipolar disorder and/or psychotic disorder)
* concurrent substance use disorder (alcohol, cannabis, stimulant, hallucinogen and/or opioid)
* using other tobacco products (electronic cigarette with nicotine, cigars or cigarillos)
* having completed an effective psychological treatment to quit smoking during the previous year
* having completed a pharmacological treatment to quit smoking in the last year (any smoking cessation medication approved by the Agencia Española del Medicamento)
* having a physical pathology involving high vital risk that requires immediate intervention (e.g., recent myocardial infarction)
* having visual difficulties that prevent the use of the App.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 429 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
7-days point prevalence abstinence | At 12-months post-intervention
  The abstinent status will be defined as not having smoked in the last 7 days (not even a puff)

SECONDARY OUTCOMES:
7-days point prevalence | At 3 and 6-months post-intervention
  The abstinent status will be defined as not having smoked in the last 7 days (not even a puff)
7-days point prevalence abstinence | At 7-days post-quit day
  The abstinent status will be defined as not having smoked in the last 7 days (not even a puff)
Satisfaction with the intervention | At 8-weeks after beginning the intervention
  Scores obtained in Client Satisfaction Questionnaire (CSQ-8; Larsen et al., 19979; Spanish version of Vázquez et al., 2017)

CONTACTS AND LOCATIONS:
Overall Officials: Ana López-Durán, Phd., Principal Investigator — University of Santiago de Compostela; Elisardo Becoña Iglesias, Phd., Principal Investigator — University of Santiago de Compostela
Locations (1):
- Smoking Cessation and Addictive Disorders Unit, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lopez-Duran A, Martinez-Vispo C, Barroso-Hurtado M, Suarez-Castro D, Becona E. Incorporating technology in smoking cessation interventions: In-person vs. Video-call formats. Int J Med Inform. 2025 Mar;195:105774. doi: 10.1016/j.ijmedinf.2024.105774. Epub 2024 Dec 24. PMID 39742855
- [Background] Martinez-Vispo C, Rodriguez-Cano R, Lopez-Duran A, Senra C, Fernandez Del Rio E, Becona E. Cognitive-behavioral treatment with behavioral activation for smoking cessation: Randomized controlled trial. PLoS One. 2019 Apr 8;14(4):e0214252. doi: 10.1371/journal.pone.0214252. eCollection 2019. PMID 30958831
- [Background] Lopez-Duran A, Martinez-Vispo C, Suarez-Castro D, Barroso-Hurtado M, Becona E. The Efficacy of the SinHumo App Combined With a Psychological Treatment to Quit Smoking: A Randomized Clinical Trial. Nicotine Tob Res. 2025 Feb 24;27(3):429-437. doi: 10.1093/ntr/ntae053. PMID 38538080
- [Background] Patnode CD, Henderson JT, Coppola EL, Melnikow J, Durbin S, Thomas RG. Interventions for Tobacco Cessation in Adults, Including Pregnant Persons: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2021 Jan 19;325(3):280-298. doi: 10.1001/jama.2020.23541. PMID 33464342